CLINICAL TRIAL: NCT05251779
Title: A Clinical Study on the Effects of Inhalation of Volatile Oil of Cang-Ai Via the Nose on Patients With Depression
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jieqiong Cui (Other)
Responsible Party: Sponsor-Investigator, Jieqiong Cui, Doctoral students, Yunnan University of Chinese Medicine
Organization: Yunnan University of Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YunnanUCM
Record Dates: First submitted 2022-01-24; First posted 2022-02-23 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Depressive Disorder; Mental Disorder in Adolescence
Keywords: Aromatic Herbs; Volatile oils; Inhalation via the nose
MeSH Terms: conditions — Depressive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cang-Ai Group (Experimental): The test group inhaled the volatile oil of Cang-Ai at a concentration of 1% by inhalation once a day for 30 minutes
  Interventions: Drug: Volatile Oil of Cang-Ai
- Bergamot group (Active Comparator): The control group inhaled the bergamot essential oils at a concentration of 1% by inhalation once a day for 30 minutes
  Interventions: Drug: Bergamot essential oils

INTERVENTIONS:
Drug: Volatile Oil of Cang-Ai — The test group will be given Volatile oil of Cang-Ai (hereafter referred to as CAVO) for inhalation
  Other Names: CAVO
  Arms: Cang-Ai Group
Drug: Bergamot essential oils — The control group will be given Bergamot essential oils for inhalation.
  Other Names: Citrus bergamia
  Arms: Bergamot group

SUMMARY:
In this study, 60 depressed patients who meet the criteria will randomly be divided into a test group and a control group, with 30 patients in each group. The test group will be given Volatile oil of Cang-Ai (hereafter referred to as CAVO) for inhalation and the control group will be given Bergamot for inhalation. The observation indicators are that after one and two sessions of the intervention, the patients' blood pressure, heart rate, depression scale scores, and changes in functional near-infrared spectroscopy(fNIRS). This randomized controlled trial will be used to look at the clinical efficacy of CAVO in patients with depression.

DETAILED DESCRIPTION:
Depression is a common psychiatric disorder characterised by persistent depressed mood, loss of interest and feelings of helplessness. Depression has the highest burden of illness of any mental illness and is the leading cause of disability. Currently, depression is usually treated with antidepressants as the first line of treatment, but because the pathophysiological mechanisms of depression are still unclear, the mechanisms of antidepressant treatment are unknown, and there is no objective way to predict efficacy, depression often requires multiple "trial and error treatments" before an effective treatment plan can be determined. Chemically synthesised drugs are widely used to treat depression, but side effects have become a bottleneck to their long-term use. As a result, natural products from medicinal plants, such as Essential oils or Volatile oils, have become research targets for the development of new drugs. Volatile oil of Cang-Ai is a component extracted from aromatic Chinese herbs such as Atractlodis Rhizoma, Herba Agastaches, Flos Caryophylli, which is commonly used clinically in the treatment of mood disorders. This study will use a randomised controlled study method. 60 patients with depression who attended the First Affiliated Hospital of Yunnan University of Traditional Chinese Medicine from March 2022 to September 2022 will be recruited.

They will be randomly divided into a trial group and a control group, 30 patients in each group. The test group will be given Volatile oil of Cang-Ai for inhalation and the control group will be given Bergamot for inhalation. Ultimately, a number of indicators will be tested to assess the clinical efficacy of the volatile oil of Cang-Ai.

ELIGIBILITY:
Inclusion Criteria:

* Meeting the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria for depressive episodes.

  * Beck Depression Scale >10; 24-item Hamilton Depression Scale (HAMD) score >20

    * Healthy sense of smell, no allergic diseases, respiratory diseases, age 16-40 years, male or female.

      * No use of antidepressants and other psychiatric drugs or physiotherapy such as electroconvulsive shock or transcranial magnetic stimulation (TMS) for at least 1 week prior to the intervention ⑤All subjects volunteered to participate and signed an informed consent form after approval by the hospital's ethics committee

Exclusion Criteria:

* History of schizophrenia, alcohol and drug dependence strictly excluded ②Depression with a history of organic brain disease and endocrine disorders or secondary to other psychiatric disorders

  * Score >3 on the Hamilton Depression Inventory for Suicide ④Pregnant and breastfeeding women with a history of manic or hypomanic episodes ⑤Family history of monophasic or bipolar disorder

Ages: 6 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from functional near-infrared spectroscopy（fNIRS) at 28 days | At the end of Cycle 1 (each cycle is 14 days)
  Functional near-infrared spectroscopy to measure changes in the relative concentrations of Oxy-Hb and Deoxy-Hb in the cerebral cortex (prefrontal and temporal lobes)
Change from functional near-infrared spectroscopy（fNIRS) at 28 days | At the end of Cycle 2 (each cycle is 14 days)
  Functional near-infrared spectroscopy to measure changes in the relative concentrations of Oxy-Hb and Deoxy-Hb in the cerebral cortex (prefrontal and temporal lobes)
24-item Hamilton Depression Inventory scores | At the end of Cycle 1 (each cycle is 14 days)
  The following severity ranges for the HAMD: no depression (0-7); mild depression (8-16); moderate depression (17-23); and severe depression (≥24)
24-item Hamilton Depression Inventory scores | At the end of Cycle 2 (each cycle is 14 days)
  The following severity ranges for the HAMD: no depression (0-7); mild depression (8-16); moderate depression (17-23); and severe depression (≥24)

SECONDARY OUTCOMES:
Change from blood pressure | At the end of Cycle 1 (each cycle is 14 days)
  Patients' blood pressure will be measured by a blood pressure monitor
Change from blood pressure at 28 days | At the end of Cycle 2 (each cycle is 14 days)
  Patients' blood pressure will be measured by a blood pressure monitor
Change from heart rate | At the end of Cycle 1 (each cycle is 14 days)
  Patients' heart rate will be measured by a heart rate monitor
Change from heart rate at 28 days | At the end of Cycle 2 (each cycle is 14 days)
  Patients' heart rate will be measured by a heart rate monitor

IPD SHARING:
Plan to Share IPD: Yes
The original data from each eligible study. including de-identified demographic information for each participant such as age, sex, nature of their health condition, as well as information about treatments or tests received and outcomes observed
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Dec 2022
Access Criteria: Sharing with researcher for Meta-analysis